CLINICAL TRIAL: NCT04497818
Title: Correlation of Fear of COVID-19 Infection and Dental Treatment Anxiety Among Netizens: A Cross-sectional Study.
Brief Title: Correlation Fear of COVID-19 & Dental Treatment Anxiety
Status: Completed | Type: Observational
Sponsor: Qassim University (Other)
Responsible Party: Principal Investigator, Dr Shiva Shankar Bugude, Assistant Professor, Qassim University
Other Study IDs: QassimU2
Record Dates: First submitted 2020-08-01; First posted 2020-08-04 (Actual); Last update posted 2020-08-04 (Actual); Status verified 2020-08

CONDITIONS: Covid19; Fear; Dental Anxiety
Keywords: Fear of COVID-19 scale; COVID-19; Modified Dental anxiety scale; Aerosols; Netizens
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Netizens: Netizens of Al Qassim province of Saudi Arabia were the target population for this cross sectional study. Sample size is (n=385) estimated based on the population size in Al Qassim province (Confidence Interval 95%, Design effect 1 & hypothesized % frequency of outcome factor of 50%). Assessment of Fear of COVID-19 was estimated using FEAR OF COVID-19, a 5 item Likert Scale. Assessment of Dental Anxiety was estimated using Modified Dental Anxiety 5 item Likert Scale. An online Survey form (Arabic 7 English) was developed using Google form application. The Google form link was shared to the netizens of Al Qassim province, across all relevant Social media platforms. Statistical analysis is done using SPSS 22.00 software program.
  Interventions: Other: Cross Sectional study using scientifically validated psychometric Scales

INTERVENTIONS:
Other: Cross Sectional study using scientifically validated psychometric Scales — Cross Sectional study using scientifically validated psychometric Scales (FEAR OF COVID-19, a 5 item Likert Scale & Modified Dental Anxiety 5 item Likert Scale).

SUMMARY:
Purpose:

COVID-19 Pandemic has created fears, anxiety and worries among general population. COVID-19 airborne transmission is possible under circumstances in which procedures generate aerosols. Various dental treatment procedures can generate aerosols. This Cross Sectional Observational study was conducted with the following objectives: 1. Assessment of Fear of COVID-19 among netizens in Al Qassim province using FEAR OF COVID-19, a 5 item Likert Scale. 2. Assessment of Dental Anxiety among netizens in Al Qassim provincen using (MDA) Modified Dental Anxiety 5 item Likert Scale.

Methods: Sample size was (n=385) estimated based on the population size in Al Qassim province (Confidence Interval 95%, Design effect 1 & hypothesized % frequency of outcome factor of 50%). Assessment of Fear of COVID-19 was estimated using FEAR OF COVID-19, a 5 item Likert Scale. Assessment of Dental Anxiety was estimated using Modified Dental Anxiety 5 item Likert Scale. An online Survey form (Arabic & English) was developed using Google form application. The Google form link was shared to the netizens of Al Qassim province, across Social media platforms. Statistical analysis is done using SPSS 22.00 software program.

DETAILED DESCRIPTION:
COVID-19 Infection was characterized as a Pandemic by WHO on the 11th of March 2020. After this there were all possible worldwide efforts to increase awareness in the general population about the COVID-19 Infection signs, symptoms, mode of transmission and prevention. The information was spread across all possible mass media communication channels.

There were constant updates regarding the data of newly infected cases, deaths, and recoveries. COVID-19 Pandemic has created fears, anxiety, and worries among the general population. COVID-19 spreads from person to person through Droplet transmission within 1-meter distance. COVID-19 airborne transmission is possible under specific circumstances and settings in which procedures or support treatments that generate aerosols. Various dental treatment procedures involve the use of equipment that can generate aerosols. Aerosols contain microorganisms and remain suspended in air in the work environment. This can potentially transfer the infectious microorganisms to the working staff and/or subsequent patients attending the Dental clinics. After the advent of COVID-19 Pandemic, there is a clear paradigm shift in Healthcare services. As the Pandemic transmission is easily transmitted through droplets and aerosols, concern regarding Dental treatment has remained as an issue.

Several past cross-sectional studies have established that Dental seeking behaviour of patients is influenced by Fear and Anxiety to Dental treatment procedures.

As the world faces COVID-19 Pandemic, the Fear of COVID-19 infection and awareness regarding COVID-19 infection can majorly influence the Dental treatment seeking behavior. General population awareness regarding droplet transmission of COVID-19 can potentially influence the fear, worry, and anxiety in Dental treatment seeking patients. The research regarding the correlation of Fear of COVID-19 to Dental treatment Anxiety is very sparse.

The psychological aspects of COVID-19 Fear and Dental anxiety have to be considered and researched.

This online Observational Cross-sectional survey study was conducted among netizens in Al Qassim province of Saudi Arabia with the following objectives:

1. To assess Fear of COVID-19 among netizins in Al Qassim province using FEAR OF COVID-19, a 5 item Likert Scale.
2. To assess Dental Anxiety among netizins in Al Qassim province using (MDA) Modified Dental Anxiety 5 item Likert Scale.
3. Correlation of Fear of COVID-19 with Dental Anxiety among Netizens in Al Qassim province.
4. Association of nearest Dental treatment seeking time and Fear of COVID.
5. Association of nearest Dental treatment seeking time and MDA.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female Human volunteer internet users who belong &/or reside in Al Qassim province region of Saudi Arabia.
* Volunteers should be major by age (18 years and above).
* People who took Dental treatment earlier in their lifetime.
* People who may take the Dental treatment in near few days or weeks or months or in a year.

Exclusion Criteria:

* Minor age group (<18 years) subjects are excluded from the study.
* Internet users who have preexisting phobia and/or anxiety mental conditions are excluded from the study.
* Internet users who are currently under treatment for their preexisting phobia and/or anxiety mental conditions are excluded from the study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Male and Female Human volunteer internet users who belong &/or reside in Al Qassim province region of Saudi Arabia are the target population for this Cross sectional study. The study population belonged to the major age group. The google form questionnaire soght for the respondents compulsory declaration of age and sound mental status. The google form also sought for the respondents compulsory consent for the survey.
Sampling Method: Probability Sample
Enrollment: 385 (Actual)
Dates: Start 2020-06-16 (Actual); Primary Completion 2020-07-16 (Actual); Study Completion 2020-07-25 (Actual)

PRIMARY OUTCOMES:
Fear of COVID-19 infection | 5th August 2020
  Assessed Fear of COVID-19 among netizens in Al Qassim province using FEAR OF COVID-19, a 5 item Likert Scale. Descriptive statistics is used to present the data.
Dental Anxiety | 5th August 2020
  Assessed Dental Anxiety among netizens in Al Qassim province using (MDA) Modified Dental Anxiety 5 item Likert Scale. Descriptive statistics is used to present the data.
Correlation of Fear of COVID-19 infection & Dental Anxiety | 5th August 2020
  The survey data is statistically analyzed to check for the correlation of the Fear of COVID-19 with Dental Anxiety among Netizens in Qassim region. The data obtained from the survey is subjected to appropriate analytical statistical tests to understand the correlation. A p-value of <0.05 is considered statistically significant correlation of the variables analysed.

SECONDARY OUTCOMES:
Correlation of the nearest Dental treatment seeking time and Fear of COVID-19 infection. | 5th August 2020
  The survey data is statistically analyzed to check for the correlation of the nearest Dental treatment seeking time and Fear of COVID-19 infection. The data obtained from the survey is subjected to appropriate analytical statistical tests to understand the correlation. A p-value of <0.05 is considered statistically significant correlation of the variables analysed.
Correlation of the nearest Dental treatment seeking time and Dental Anxiety | 5th August 2020
  The survey data is statistically analyzed to check for the correlation of the nearest Dental treatment seeking time and Dental Anxiety. The data obtained from the survey is subjected to appropriate analytical statistical tests to understand the correlation. A p-value of <0.05 is considered statistically significant correlation of the variables analysed.
Correlation of the Age and Fear of COVID-19 infection | 5th August 2020
  The survey data is statistically analyzed to check for the correlation of Age and Fear of COVID-19 infection The data obtained from the survey is subjected to appropriate analytical statistical tests to understand the correlation. A p-value of <0.05 will be considered statistically significant correlation of the variables analysed.
Correlation of the Age and Dental Anxiety. | 5th August 2020
  The survey data is statistically analyzed to check for the correlation of the Age and Dental Anxiety. The data obtained from the survey is subjected to appropriate analytical statistical tests to understand the correlation. A p-value of <0.05 is considered statistically significant correlation of the variables analysed.

CONTACTS AND LOCATIONS:
Overall Officials: Bugude Shiva Shankar, Principal Investigator — College of Applied Health Sciences - Al Rass
Locations (1):
- Dr Bugude Shiva Shankar, Ar Rass, Al Qassim, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided
The Research data will be available to the Principal Investigator. On requirement the data will be shared to whomsoever after consultation with the concerned higher authorities in the College of Applied Health sciences in Ar rass. The descriptive & analytical data will be used for scientific publication.